CLINICAL TRIAL: NCT07395687
Title: A Study Investigating Safety, Tolerability and Efficacy of UBT251 in Participants Living With Overweight or Obesity
Brief Title: A Research Study on How Well Different Doses of the Medicine UBT251 Help People Living With Overweight or Obesity
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9559-8568; U1111-1324-3831 (Other: World Health Organization (WHO))
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part A - UBT251 (Experimental): Participants will be randomized to receive multiple dose levels subcutaneously.
  Interventions: Drug: UBT251
- Part A - placebo (Placebo Comparator): Participants will receive placebo matched to UBT251 subcutaneously.
  Interventions: Drug: Placebo
- Part B - Arm A (UBT251) (Experimental): Participants will be randomized to receive multiple dose levels subcutaneously.
  Interventions: Drug: UBT251
- Part B - Arm B (UBT251) (Experimental): Participants will be randomized to receive multiple dose levels subcutaneously.
  Interventions: Drug: UBT251
- Part B - Arm C (UBT251) (Experimental): Participants will be randomized to receive multiple dose levels subcutaneously.
  Interventions: Drug: UBT251
- Part B - Arm D (UBT251) (Experimental): Participants will be randomized to receive 2 dose levels subcutaneously.
  Interventions: Drug: UBT251
- Part B - Arm E (UBT251) (Experimental): Participants will be randomized to receive a single dose level subcutaneously.
  Interventions: Drug: UBT251
- Part B - placebo (Placebo Comparator): Participants will receive placebo matching one of the UBT251 arms subcutaneously.
  Interventions: Drug: Placebo
- Part C - UBT251 dose 1 (Experimental): Participants will be randomized to receive dose level 1 subcutaneously.
  Interventions: Drug: UBT251
- Part C - UBT251 dose 2 (Experimental): Participants will be randomized to receive dose level 2 subcutaneously.
  Interventions: Drug: UBT251
- Part C - UBT251 dose 3 (Experimental): Participants will be randomized to receive dose level 3 subcutaneously.
  Interventions: Drug: UBT251

INTERVENTIONS:
Drug: UBT251 — UBT251 injection will be administered subcutaneously in a lifted fold of the abdominal skin.
  Arms: Part A - UBT251; Part B - Arm A (UBT251); Part B - Arm B (UBT251); Part B - Arm C (UBT251); Part B - Arm D (UBT251); Part B - Arm E (UBT251); Part C - UBT251 dose 1; Part C - UBT251 dose 2; Part C - UBT251 dose 3
Drug: Placebo — Placebo matched to UBT251 injection will be administered subcutaneously in a lifted fold of the abdominal skin.
  Arms: Part A - placebo; Part B - placebo

SUMMARY:
The purpose of this clinical study is to find out if UBT251 is safe and effective for treating people who are living with overweight or obesity. Participants will get either UBT251 (the treatment being tested) or Placebo (a treatment that has no active medicine in it), which treatment participants get is decided by chance.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (sex at birth).
2. For Part C: Japanese, Chinese or non-Asian participants (all self-reported):

   * For Japanese participants: both parents of Japanese descent.
   * For Chinese participants: both parents of Chinese descent.
   * For non-Asian participants: both parents of non-Asian descent (non-Asian is defined as of countries outside of Asia).
3. Age at the time of signing the informed consent:

   1. For Part A: 18-55 years (both inclusive)
   2. For Part B: 18-65 years (both inclusive)
   3. For Part C: 18-55 years (both inclusive).
4. BMI at screening (overweight and obesity should be due to excess adipose tissue, as judged by the investigator):

   1. For Part A: 27.0-39.9 kilogram per meter square (kg/m^2) (both inclusive)
   2. For Part B: 30.0-50.0 kg/m^2 (both inclusive)
   3. For Part C: 24-34.9 kg/m^2 (both inclusive)
5. Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG), and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

1. Known or suspected hypersensitivity to study intervention(s) or related products.
2. Treatment with any marketed product containing compounds with glucagon-like peptide 1 (GLP-1), glucose-dependent insulinotropic polypeptide (GIP) or glucagon receptor agonism within 90 days before screening.
3. Any condition, unwillingness or inability, which in the investigator's opinion might jeopardise the participant's safety or compliance with the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-01-14 (Estimated); Study Completion 2027-02-18 (Estimated)

PRIMARY OUTCOMES:
Part A - Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to end of study (week 33)
  Measured as Number of events.
Part B - Relative change in body weight | From baseline (week 0) to end of treatment (week 28)
  Measured as percentage of body weight.
Part C- AUC; the area under the UBT251 plasma concentration time curve | From pre-dose on Day 1 until completion of the end of study visit (Day 43)
  Measured as hour*nanomoles per liter (h*nmol/L)

SECONDARY OUTCOMES:
Part A - Relative change in body weight | From baseline (week 0) to end of treatment (week 28)
  Measured as percentage of body weight.
Part A - Change in body weight | From baseline (week 0) to end of treatment (week 28)
  Measured as kilogram (kg).
Part A - AUC; the area under the UBT251 plasma concentration-time curve | From pre-dose on day 1 to end of study (week 33)
  Measured as h*nmol/L
Part A - Cmax; the maximum plasma concentration of UBT251 | From pre-dose on day 1 to end of study (week 33)
  Measured as nanomole per liter (nmol/L)
Part B - Change in body weight | From baseline (week 0) to end of treatment (week 28)
  Measured as kg.
Part B - Change in waist circumference | From baseline (week 0) to end of treatment (week 28)
  Measured as centimetre (cm).
Part B - Number of TEAEs | From baseline (week 0) to end of study (week 33)
  Measured as number of events
Part C - Cmax; the maximum plasma concentration of UBT251 | From pre-dose on Day 1 until completion of the end of study visit (Day 43)
  Measured as nmol/L
Part C - Number of treatment-emergent adverse events (TEAEs) | From pre-dose on Day 1 until completion of the end of study visit (Day 43)
  Measured as number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (3):
- United States (2):
  - Altasciences Clinical LA, Inc., Cypress, California
  - Altasciences Clinical Kansas, Inc., Overland Park, Kansas
- Altasciences Clinical Company, Inc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com